CLINICAL TRIAL: NCT03922672
Title: The Impact of Group Piano Training on Psychosocial Outcomes in Caregivers of Adults With Parkinson's Disease
Brief Title: Piano Training, Caregivers, and Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Teresa Lesiuk, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180888
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Depression; Mood; Burden, Dependency
Keywords: caregiver; Parkinson's disease; group piano training
MeSH Terms: conditions — Depression; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Piano group (Experimental): This group will consist of the adult with Parkinson's disease and their caregiver for a total of 14 pairs.
  Interventions: Behavioral: Group piano training

INTERVENTIONS:
Behavioral: Group piano training — The group piano training is scheduled over 4 months of a two-hour weekly group piano lesson. There is also a 3-hour weekly practice at home.

SUMMARY:
The purpose of this study is to investigate the impact of group piano training on psychosocial outcomes in caregivers of adults with Parkinson's disease (PD). As well, the study is investigating the impact of group piano training on psychosocial outcomes in the care-recipient with PD.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver:

  * Are currently a primary caregiver to an adult with PD
  * Are between the age of 40-80 years
  * Have less than 5 years of music training
  * Speak and read English fluently

Adult with PD:

* Stage 1-3 Parkinson's disease
* Are between the age of 40-80
* Have less than 5 years of music training
* Speak and read English fluently

Exclusion Criteria:

* Doesn't meet all the inclusion criteria

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Change in caregiver burden as assessed by the Zarit Burden Interview. | Baseline to month 1, baseline to month 2, baseline to month 4
  The Zarit burden is a 22-item questionnaire with range from 0-88 with a higher score indicating severe burden.

SECONDARY OUTCOMES:
Change in depression as assessed by the Center for Epidemiological Studies for Depression (CES-D). | Baseline to month 1, baseline to month 2, baseline to month 4
  The CES-D is a 20-item questionnaire with range from 0-60 with a higher score indicating increased symptoms of depression.
Change in musical self-efficacy as assessed by the Musical Performance Self-Efficacy Scale (MPSE). | Baseline to month 1, baseline to month 2, baseline to month 4
  The MPSE is a 24 item questionnaire with range from 0-2400 with a higher score indicating improved musical self-efficacy.
Change in mood by the Profile of Mood States - Brief Form (POMS-BF). | From month 1 to month 4.
  The POMS-BF is a 30 item questionnaire with six sub-scale scored on a 5-point Likert scale with a higher total score indicating increased negative mood.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa L Lesiuk, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No